CLINICAL TRIAL: NCT06825897
Title: Delay Avoiding Primary Evaluation for Thrombectomy for Acute Stroke Patients With Large Vessel Occlusion in the Angiography Suite (DIRECT) Trial
Brief Title: Delay AvoIding Primary Evaluation for ThRombectomy of Acute StrokE Patients With Large Vessel OCclusion in the Angiography SuiTe
Acronym: DIRECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Santiago Ortega Gutierrez (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Santiago Ortega Gutierrez, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202407139
Record Dates: First submitted 2025-01-29; First posted 2025-02-13 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Stroke, Acute
Keywords: Large Vessel Occlusion; Acute Ischemic Stroke; Pragmatic Clinical Trial
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This study employs a cluster-randomized crossover design, where thrombectomy-capable stroke centers (clusters) are randomized to adopt one of two standard-of-care triage strategies: direct transfer to the neurointerventional angiography suite or conventional emergency department evaluation. Each cluster transitions between strategies at predefined intervals of two weeks. This design ensures all centers implement both approaches, enabling a robust comparison of clinical outcomes while accommodating site-specific workflows and variability.
Who Masked: Participant, Outcomes Assessor
Masking Description: Data Analysts: Individuals analyzing the data may also be blinded to the treatment assignment to avoid bias in data interpretation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Triage Arm (Active Comparator): In this arm, patients with suspected large vessel occlusion (LVO) stroke undergo an initial evaluation in the emergency department (ED), including standard imaging, to confirm eligibility for mechanical thrombectomy (MT). Once eligibility is confirmed, they are transferred to the neurointerventional suite for further treatment. This strategy represents the traditional approach used in many stroke centers and serves as a comparator to the direct transfer strategy. The outcomes measured in this arm will be compared to those in the Direct Transfer to Angiography Suite (DTAS) arm to assess the relative effectiveness and safety of both triage strategies.
  Interventions: Other: Conventional Triage for Mechanical Thrombectomy
- Direct Transfer to Angiography Suite (DTAS) Arm (Active Comparator): Description: In this arm, patients with suspected large vessel occlusion (LVO) stroke are directly transferred to the neurointerventional angiography suite without initial evaluation in the emergency department. Neuroimaging is performed using flat panel CT (FPCT) to confirm treatment eligibility for mechanical thrombectomy (MT). This strategy aims to reduce delays in treatment and improve clinical outcomes by bypassing the emergency department, leading to faster access to thrombectomy. This arm will assess the effectiveness and safety of direct transfer, comparing it to the conventional triage strategy in terms of disability outcomes, safety, and healthcare utilization.
  Interventions: Other: Direct Transfer to Angiography Suite (DTAS

INTERVENTIONS:
Other: Conventional Triage for Mechanical Thrombectomy — Participants undergo the conventional standard-of-care triage process. Upon arrival at the thrombectomy-capable center, patients first undergo an initial evaluation in the emergency department (ED), which includes diagnostic imaging (CT or MRI) to confirm eligibility for mechanical thrombectomy (MT). If the patient is found to have a large vessel occlusion (LVO) suitable for thrombectomy, they are transferred to the neurointerventional suite for treatment.
  Arms: Conventional Triage Arm
Other: Direct Transfer to Angiography Suite (DTAS — Patients who arrive at the thrombectomy-capable center (from home, mobile stroke units, or interfacility transfer) are immediately transferred to the neurointerventional suite, bypassing the emergency department (ED). Upon arrival in the neurointerventional suite, initial neuroimaging (typically using flat panel CT or other imaging modalities) is conducted to confirm the presence of a large vessel occlusion (LVO). If the patient is eligible for mechanical thrombectomy (MT), treatment is initiated directly in the angiography suite. This approach aims to reduce delays in care and improve clinical outcomes by providing faster access to thrombectomy treatment.
  Arms: Direct Transfer to Angiography Suite (DTAS) Arm

SUMMARY:
The purpose of this study is to compare two strategies for treating adults with suspected large vessel occlusion stroke within 7 hours of symptom onset. Researchers will evaluate whether direct transfer to the neurointerventional angiography suite improves recovery and reduces disability compared to the conventional approach of first being evaluated in the emergency department. The study will also assess safety and other health outcomes to guide care for stroke patients.

DETAILED DESCRIPTION:
Large vessel occlusion (LVO) strokes are among the most severe types of strokes, caused by a blockage in one of the brain's major blood vessels. These strokes can lead to significant disability or death without prompt treatment. Mechanical thrombectomy (MT), a procedure that physically removes the clot, is one of the most effective treatments for LVO strokes. However, there is still uncertainty about the best way to quickly triage and prepare patients for MT to achieve the best outcomes.

This study, called the DIRECT trial, aims to compare two common triage strategies for patients suspected of having an LVO stroke:

Direct transfer to the neurointerventional angiography suite - In this strategy, patients are taken straight to the neurointerventional suite upon arrival at the hospital. Advanced imaging and treatment decisions are made immediately, potentially speeding up treatment.

Conventional evaluation in the emergency department (ED) - In this approach, patients undergo initial evaluation and imaging in the ED before being transferred to the neurointerventional suite if they are eligible for MT.

The main goal of this study is to determine if bypassing the ED and directly transferring patients to the neurointerventional suite leads to better recovery and reduced disability at 90 days compared to the conventional strategy. Researchers will also assess other important outcomes, including safety (such as the risk of brain bleeding), quality of life after the stroke, efficiency of stroke care, and the use of healthcare resources (such as hospital stay length).

The study will include approximately 2,039 adult patients aged 18 and older who are suspected of having an LVO stroke. To participate, patients must arrive at one of the participating thrombectomy-capable stroke centers within 7 hours of symptom onset. These centers are equipped to perform advanced stroke care, including MT.

Participants in the trial will represent a diverse population reflective of the general community affected by stroke. The trial will take place at 20 hospitals across the United States, all with high experience in treating stroke patients. The study will help provide critical insights into which triage strategy offers the best outcomes for patients with LVO strokes and improve future care for these emergencies.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in the DIRECT trial, an individual must meet all of the following criteria:

1. Age: ≥ 18 years of age.
2. Clinical Presentation: Present to a participating TSC with signs or symptoms suggestive of acute LVO stroke.
3. Stroke Severity: Baseline NIHSS of 10 or higher.
4. Time since LKW: Time from LKW to arrival at the TSC must be within 7 hours.

Additional criteria

For all Interfacility Transfers:

1. If imaging was performed at the outside facility, the time from the first imaging to arrival at the thrombectomy center must exceed 90 minutes.

For all the Conventional Triage Arm, participants must also meet the following criteria:

1. Presence of a qualifying LVO by CTA or MRA imaging; or
2. For Large Core Patients: Patients with large core infarcts (CT-ASPECT score ≤ 5, DWI-ASPECT score ≤ 5, or infarct volume ≥ 70 cc) will be enrolled, irrespective of treatment decisions regarding embolectomy.

For all DTAS Arm:

1. Patients who do not have LVO occlusions in the angiography suite assessment (ICH, distal occlusions or mimics) will be enrolled, irrespective of treatment decisions regarding embolectomy.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in the trial:

1. Time Restrictions: Presentation to a thrombectomy-capable center more than 7 hours from LSW.
2. Imaging Criteria for Interfacility Transfer Patients: At sites enrolling transfer patients, any patient arriving from an outside hospital with time from imaging study at the presenting hospital to arrival at the TSC not exceeding 90 minutes.
3. Hemorrhagic Stroke: Presence of intracranial hemorrhage on brain imaging in the conventional strategy as Heidelberg that renders thrombectomy contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2039 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Global Disability at 90 Days | 90 days (±14 days)
  Global disability will be measured using the disability-weighted modified Rankin Scale (dw-mRS) at 90 days (±14 days) post-stroke. The dw-mRS is a validated tool assessing the severity of disability across seven levels, from no symptoms (0) to severe disability or death (6). This outcome evaluates whether the direct transfer to the angiography suite (DTAS) strategy results in improved functional outcomes compared to the conventional triage strategy.

SECONDARY OUTCOMES:
Functional Independence at 90 Days | 90 (±14) days.
  The proportion of patients achieving functional independence, measured by a dichotomized modified Rankin Scale score (mRS 0-2), assessed during the in-hospital stay and at 90 (±14) days after treatment.
Stroke Workflow Efficiency | Immediately post procedure
  Metrics include door-to-puncture times, door-to-reperfusion times, and rates of intravenous thrombolysis administration, evaluating the time taken to perform key steps in stroke workflow.
Procedural Success | Immediately post-procedure.
  Reperfusion rates of the large vessel occlusion (LVO) using the Extended Thrombolysis in Cerebral Ischemia (eTICI) scale, with successful reperfusion defined as mTICI 2b-3.
Cognitive Ability | 90 (±14) days.
  Assessed at 90 days using the Montreal Cognitive Assessment (MoCA), measuring domains such as memory, attention, and executive function.
Health-Related Quality of Life | 90 (±14) days.
  HR-QoL evaluated using PROMIS GH-10 and EQ-5D-5L to assess overall health and well-being at 90 days.

OTHER OUTCOMES:
Global Disability | Immediately at discharge.
  Disability measured by all seven ordinal levels of the modified Rankin Scale (mRS) at hospital discharge.
Instrumental Activities of Daily Living | 90 (±14) days.
  Measured at 90 days using the Barthel Index, assessing the patient's ability to perform daily activities independently.
Caregiving Burden | 90 (±14) days.
  Caregiving burden assessed using Zarit's Burden Interview (ZBI) at 90 days, evaluating the impact of stroke on caregivers.
Healthcare Utilization | 90 (±14) days.
  Assessed by metrics such as length of hospital stay, home-time, and number of days spent at initial residency level within 90 days post-stroke.
Mortality | 90 (±14) days.
  Mortality rates assessed at 90 days and during the in-hospital stay.
Procedural Complications | Immediately post procedure
  Intraprocedural complications such as vessel perforation, arterial dissection, access site complications, and intraprocedural mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Ortega, MD, Principal Investigator — University of Iowa; Tudor Jovin, MD, Principal Investigator — Cooper University Health Care
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] Galecio-Castillo M, Vivanco-Suarez J, Zevallos CB, Dajles A, Weng J, Farooqui M, Ribo M, Jovin TG, Ortega-Gutierrez S. Direct to angiosuite strategy versus standard workflow triage for endovascular therapy: systematic review and meta-analysis. J Neurointerv Surg. 2023 Sep;15(e1):e17-e25. doi: 10.1136/neurintsurg-2022-018895. Epub 2022 Jun 16. PMID 35710313
- [Background] Nogueira RG, Jadhav AP, Haussen DC, Bonafe A, Budzik RF, Bhuva P, Yavagal DR, Ribo M, Cognard C, Hanel RA, Sila CA, Hassan AE, Millan M, Levy EI, Mitchell P, Chen M, English JD, Shah QA, Silver FL, Pereira VM, Mehta BP, Baxter BW, Abraham MG, Cardona P, Veznedaroglu E, Hellinger FR, Feng L, Kirmani JF, Lopes DK, Jankowitz BT, Frankel MR, Costalat V, Vora NA, Yoo AJ, Malik AM, Furlan AJ, Rubiera M, Aghaebrahim A, Olivot JM, Tekle WG, Shields R, Graves T, Lewis RJ, Smith WS, Liebeskind DS, Saver JL, Jovin TG; DAWN Trial Investigators. Thrombectomy 6 to 24 Hours after Stroke with a Mismatch between Deficit and Infarct. N Engl J Med. 2018 Jan 4;378(1):11-21. doi: 10.1056/NEJMoa1706442. Epub 2017 Nov 11. PMID 29129157
- [Background] Regenhardt RW, Rosenthal JA, Dmytriw AA, Vranic JE, Bonkhoff AK, Bretzner M, Hirsch JA, Rabinov JD, Stapleton CJ, Patel AB, Singhal AB, Rost NS, Leslie-Mazwi TM, Etherton MR. Direct to angio-suite large vessel occlusion transfers achieve faster arrival-to-puncture times and improved outcomes. Stroke Vasc Interv Neurol. 2022 Nov;2(6):e000327. doi: 10.1161/svin.121.000327. Epub 2022 Jul 5. PMID 36571077
- [Background] Mendez B, Requena M, Aires A, Martins N, Boned S, Rubiera M, Tomasello A, Coscojuela P, Muchada M, Rodriguez-Luna D, Rodriguez-Villatoro N, Juega J, Pagola J, Molina CA, Ribo M. Direct Transfer to Angio-Suite to Reduce Workflow Times and Increase Favorable Clinical Outcome. Stroke. 2018 Nov;49(11):2723-2727. doi: 10.1161/STROKEAHA.118.021989. PMID 30355182
- [Background] Ribo M, Boned S, Rubiera M, Tomasello A, Coscojuela P, Hernandez D, Pagola J, Juega J, Rodriguez N, Muchada M, Rodriguez-Luna D, Molina CA. Direct transfer to angiosuite to reduce door-to-puncture time in thrombectomy for acute stroke. J Neurointerv Surg. 2018 Mar;10(3):221-224. doi: 10.1136/neurintsurg-2017-013038. Epub 2017 Apr 26. PMID 28446535
- [Background] Almekhlafi MA, Goyal M, Dippel DWJ, Majoie CBLM, Campbell BCV, Muir KW, Demchuk AM, Bracard S, Guillemin F, Jovin TG, Mitchell P, White P, Hill MD, Brown S, Saver JL; HERMES Trialists Collaboration. Healthy Life-Year Costs of Treatment Speed From Arrival to Endovascular Thrombectomy in Patients With Ischemic Stroke: A Meta-analysis of Individual Patient Data From 7 Randomized Clinical Trials. JAMA Neurol. 2021 Jun 1;78(6):709-717. doi: 10.1001/jamaneurol.2021.1055. PMID 33938914
- [Background] Ribo M, Alvarez-Sabin J, Montaner J, Romero F, Delgado P, Rubiera M, Delgado-Mederos R, Molina CA. Temporal profile of recanalization after intravenous tissue plasminogen activator: selecting patients for rescue reperfusion techniques. Stroke. 2006 Apr;37(4):1000-4. doi: 10.1161/01.STR.0000206443.96112.d9. Epub 2006 Mar 2. PMID 16514102
- [Background] Jovin TG, Li C, Wu L, Wu C, Chen J, Jiang C, Shi Z, Gao Z, Song C, Chen W, Peng Y, Yao C, Wei M, Li T, Wei L, Xiao G, Yang H, Ren M, Duan J, Liu X, Yang Q, Liu Y, Zhu Q, Shi W, Zhu Q, Li X, Guo Z, Yang Q, Hou C, Zhao W, Ma Q, Zhang Y, Jiao L, Zhang H, Liebeskind DS, Liang H, Jadhav AP, Wen C, Brown S, Zhu L, Ye H, Ribo M, Chang M, Song H, Chen J, Ji X; BAOCHE Investigators. Trial of Thrombectomy 6 to 24 Hours after Stroke Due to Basilar-Artery Occlusion. N Engl J Med. 2022 Oct 13;387(15):1373-1384. doi: 10.1056/NEJMoa2207576. PMID 36239645
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510